CLINICAL TRIAL: NCT02124603
Title: Evaluation of Ocular Flora in Patients Undergoing Cataract Surgery. An Observational Study
Brief Title: Microbiological Evaluation of the Ocular Flora Before Cataract Surgery
Status: Completed | Type: Observational
Sponsor: SIFI SpA (Industry)
Responsible Party: Sponsor
Other Study IDs: 041SI
Record Dates: First submitted 2014-04-23; First posted 2014-04-28 (Estimated); Results first posted 2015-09-29 (Estimated); Last update posted 2016-01-18 (Estimated); Status verified 2015-12

CONDITIONS: Disorders of the Eye Following Cataract Surgery
Keywords: cataract; prophylaxis; susceptibility
MeSH Terms: conditions — Cataract; Disease Susceptibility

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Conjunctival and palpebral swab of the eye undergoing surgery
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- single group: Patients undergone cataract surgery

SUMMARY:
The purpose of the present study is to elucidate the spectrum of ocular flora and their antimicrobial susceptibility profiles in patients undergoing routine cataract surgery.

DETAILED DESCRIPTION:
A conjunctival and palpebral swab will executed at least 14 days before routine cataract surgery. Isolates will be identified using standard microbiological protocols. In vitro susceptibility will be determined using a breakpoint minimal inhibitory concentrations. In case of positivity, the swab will be repeated the day of surgery. Topical antibiotic may be used in case of positivity at the discretion of the surgeon. Descriptive statistics will be calculated.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for cataract surgery
* Age > 18 years
* Any gender and race
* Willing to sign informed consent

Exclusion Criteria:

* Any antibiotics within 3 months
* Any ocular infection within 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing routine cataract surgery
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2014-04; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marcello Santocono, MD, Principal Investigator — Casa Di Cura Di Stefano Catania (Italy)
Locations (1):
- Casa di Cura Di Stefano, Catania, Catania, Italy

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Single Group
Started | 120
Completed | 120
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Single Group: Consecutive patients scheduled for cataract surgery
Arm/Group | Single Group
Number analyzed (Participants) | 120
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.3 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 71
  Male | 49
Region of Enrollment [Number; unit: participants]
  Italy | 120

OUTCOME MEASURES:

1. Primary Outcome: Positive Culture in Subjects Scheduled for Cataract Surgery
Description: Number of participants with positive culture at the screening visit
Time Frame: At least 14 days before surgery
Population: Number of participants with positive culture
Measure: Number; unit: subjects
Arm/Group | Single Group
Number analyzed (Participants) | 120
subjects | 87

2. Secondary Outcome: Antibiotic Susceptibility
Description: Isolated bacteria were tested for their in vitro susceptibility to commercially available ophthalmic antibiotics by the disk diffusion test and categorized as susceptible, intermediate or resistant.
Time Frame: At least 14 days before surgery
Population: Percentage of isolates susceptibility to antibiotics
Measure: Number; unit: percentage of susceptible isolates
Units Other Than Participants: strains
Arm/Group | Single Group
Number analyzed (Participants) | 120
Number analyzed (strains) | 131
percentage of susceptible isolates
  netilmicin | 94
  moxifloxacin | 86
  chloramphenicol | 74
  levofloxacin | 70
  tobramycin | 59
  ofloxacin | 57
  azythromycin | 15

3. Secondary Outcome: Eradication Rate
Description: Number of participants having positive culture at the screening visit with bacterial eradication before surgery
Time Frame: Day of surgery
Population: Number of participants with positive culture at the screening visit
Measure: Number; unit: partecipants
Arm/Group | Single Group
Number analyzed (Participants) | 87
partecipants | 80

ADVERSE EVENTS:
Groups:
- Single Group: Patients to have to undergone cataract surgery
Arm/Group | Single Group
Serious Adverse Events (participants affected / at risk) | 0/120
Other Adverse Events (participants affected / at risk) | 0/120

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No